CLINICAL TRIAL: NCT04516408
Title: Efficacy and Safety of Recombinant Zoster Vaccine in Stable SLE Patients(Vtrial)
Brief Title: Recombinant Zoster Vaccine in Stable SLE Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vtrial
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Herpes Zoster; Recombinant Zoster Vaccine; Systemic Lupus Erythematosus
MeSH Terms: conditions — Herpes Zoster; Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: Herpes Zoster
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant zoster vaccine (Experimental): Eligible patients were randomized in a 1:1 ratio to recombinant zoster vaccine/placebo on the background of standard of care (SOC). Participants received two intramuscular doses of the vaccine 2 months apart.
  Interventions: Biological: Recombinant zoster vaccine
- Placebo (Placebo Comparator): Eligible patients were randomized in a 1:1 ratio to recombinant zoster vaccine/placebo on the background of standard of care (SOC). Participants received two intramuscular doses of the placebo (sterilized water) 2 months apart.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Recombinant zoster vaccine — Recombinant zoster vaccine (RZV) is indicated for prevention of herpes zoster in adults aged ≥ 50 years old. RZV contains a varicella zoster virus glycoprotein E antigen and the AS01B adjuvant system.
  Arms: Recombinant zoster vaccine
Biological: Placebo — Sterilized water
  Arms: Placebo

SUMMARY:
The risk of herpers zoster reactivation is higher in SLE patients than general population. It has shown that mild or even inactive patients could also have varicella zoster virus (VZV) infections, and they account for about two-thirds of the events. And our previous study indicated that recent various VZV infection was associated with increased risk of disease flares. The risk of virus reactivation limited the use of live-attenuated shingles vaccine in SLE patients, especially in whom with high dose of prednisone or immunosuppressants. Whether the introduction of recombinant zoster vaccine could reduce the risk of zoster reactivation in lupus patients is to be explored in this study.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic systemic autoimmune disease that requires long-term corticosteroid and/or immunosuppressive agents. Thus lupus patients are immunocompromised patients, and the incidence of herpes zoster is higher than general population (asian population 32.5-91.4/1000 person-years vs general population 2.58-4.89/1000 person-years). Patients with active SLE are more susceptible because they require stronger immunosuppressive therapy. However, even mild or even stable lupus patients are highly susceptible, and they account for about two-thirds of the events. In addition, herpes zoster may trigger lupus flare. A case-control study showed a close correlation between herpes zoster reactivation and the diagnosis of lupus, and our previous studies indicated that recent VZV infection was associated with increased risk of disease flares. The risk of virus reactivation limited the use of live-attenuated shingles vaccine in SLE patients, especially in whom with high dose of prednisone or immunosuppressants. Whether the introduction of recombinant herpes zoster could reduce the risk of zoster reactivation in lupus patients is to be explored in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years old
2. The disease status is stable (score≤ 6 at screening on SELENA-SLEDAI); no British Isles Lupus Assessment Group (BILAG) A and no more than one BILAG B;
3. A stable treatment regimen with fixed doses of prednisone (≤ 20mg/day), antimalarial, or immunosuppressive drugs (azathioprine/mycophenolate mofetil/ methotrexate/ciclosporin/tacrolimus/leflunomide/belimumab);
4. Sign the informed consent.

Exclusion Criteria:

1. Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) > 2 times upper normal limits; creatinine clearance rate < 60ml/min;
2. Exposure to cyclophosphamide within the past half year.
3. Exposure to rituximab within the past one year.
4. History of herpes zoster within the past three months;
5. Pregnancy or lactation;
6. History of malignancy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Percent of participants with herpes zoster | 12 months
  The efficacy of recombinant zoster vaccine in stable systemic lupus patients

SECONDARY OUTCOMES:
Immunogenicity | Baseline, 3 month, and 12 month
  Humoral immunity was measured as geometric mean concentrations (GMCs) of serum anti-gE antibodies (ELISA), and CMI was measured as the frequency of CD4 T cells expressing ≥ 2 of 4 selected activation markers (interferon-γ, interleukin-2, tumour necrosis factor-α and CD40 ligand) per 10^6 CD4 T cells after stimulation with gE peptides (hereafter referred to as CD4^2+ T cells)
Percent of participants with lupus flares | 12 months
  either minor/moderate flare or major flare defined by SLEDAI Flare Index
Change of interferon score during follow-up | 12 months
  Interferon score is detected at each visit, the time of herpes zoster and lupus flare.
Adverse events | 12 months
  To evaluate for adverse effects following immunization patients will submit the adverse effects by app tracking system.

CONTACTS AND LOCATIONS:
Overall Officials: Fangfang Sun, MD., Principal Investigator — Renji Hospital, Shouth Campus
Locations (1):
- Shuang Ye, MD, Shanghai, Shanghai Municipality, China